CLINICAL TRIAL: NCT00655187
Title: Case-control Study to Evaluate the Vaccine Effectiveness of Rotarix™ Against Rotavirus Severe Gastroenteritis (RV SGE) Among Hospitalised Children < 5 Years of Age in KK Hospital, Singapore
Brief Title: Effectiveness of Human Rotavirus Vaccine, Rotarix™ Against Rotavirus Severe Gastroenteritis (RV SGE) in Infants
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 110467
Record Dates: First submitted 2008-04-01; First posted 2008-04-09 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Rotavirus Severe Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples

GROUPS / COHORTS (2):
- Group A: Cases
  Interventions: Other: Collection of information; Procedure: Collection of stool samples
- Group B: Controls
  Interventions: Other: Collection of information

INTERVENTIONS:
Other: Collection of information — Information regarding demographic characteristics, medical history, previous participation in rotavirus clinical trials and vaccination history will be collected.
Procedure: Collection of stool samples — Stools samples will be collected during hospitalisation for RV testing and genotyping of RV positive samples.
  Groups: Group A

SUMMARY:
This study aims to evaluate the effectiveness of Rotarix™ vaccine in the general population in Singapore by monitoring the overall reduction in RV SGE and also by assessing the direct protection offered by the vaccine in hospitalised infants through a case-control study.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following an amendment of the Protocol.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for surveillance subjects

* A male or female child aged < 60 months at the time of admission (a child becomes ineligible on the day of its fifth birthday).
* Subject admitted with acute GE as an inpatient to the study site during the study period.
* Written informed consent obtained from the parent or guardian of the subject. Selection criteria for cases

Cases will be limited to those surveillance subjects:

* who are born after 1 November 2005 (date of availability of Rotarix™ vaccination in Singapore),
* who are aged at least 16 weeks at the time of hospital admission.
* whose stool samples are tested positive for RV. Selection criteria for controls

All controls must satisfy the following criteria at study entry:

* Admitted for acute disease with non-GE causes in the same hospital as the case , with the closest admission date to the cases.
* Aged at least 16 weeks at the time of hospital admission.
* Born within a range of ± 2 weeks from the date of birth of cases. In case there is no suitable match, then the range would be extended to ± 4 weeks.
* Written informed consent obtained from the subject's parents/guardians.

Exclusion Criteria:

For enrolment of surveillance subjects

The following criteria should be checked at the time of study entry. If any apply, the subject must not be included in the study:

* The diagnoses at admission to the study site do not include acute GE.
* Children for whom stool samples are not available up to 48 hours after admission.
* The onset of GE is after 48 hours of admission to the hospital (i.e. nosocomial GE).
* Children with a history of chronic and genetic diseases. For selection of cases

In addition to the exclusion criteria for surveillance subjects, cases will not be selected if the following criterion applies:

* Subjects who had a previous episode of acute GE less than a week back i.e. recurrent GE episode.
* Subjects who have been already enrolled in the study.
* Subjects whose vaccination history could not be ascertained. For selection of controls

The following criteria should be checked at the time of study entry. If any apply, the controls must not be included in the study:

* Child who has symptoms of GE on the day of interview of his/her parent or guardian or had an episode of GE within 14 days prior to the day of interview.
* Child who has been already enrolled in the study as case or control.
* The onset of GE occurs after admission at the hospital.
* Child whose vaccination history could not be ascertained.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children less than 5 years of age, hospitalised with acute GE, living in Singapore served by the hospital participating in the study (KK Hospital) and whose parents/ guardians are willing to provide informed consent, will be considered as cases.
  Cases will be limited to those subjects who are born after 1 November 2005, aged at least 16 weeks and whose stool samples have been tested positive for rotavirus (RV).
  For each case, two controls hospitalised for acute disease with non-GE causes in the same hospital during the same period, will be included in the study after matching them by date of birth.
Sampling Method: Probability Sample
Enrollment: 1270 (Actual)
Dates: Start 2008-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To estimate the proportion of acute RV GE hospitalisations in children < 5 years of age. | At least one year
To estimate the effectiveness of two doses of Rotarix™ vaccination in preventing rotavirus severe gastroenteritis (RV SGE) among children born after 1 November 2005 and aged at least 16 weeks. | At least one year

SECONDARY OUTCOMES:
To estimate the effectiveness of two doses of Rotarix™ vaccination in preventing hospitalisation for acute RV GE among children born after 1 November 2005 and aged at least 16 weeks. | At least one year
To determine the distributions of acute RV GE associated hospital admissions according to subject's age, gender and by month of year. | At least one year
To estimate the prevalence of RV genotypes in acute RV GE associated hospital admission. | At least one year
To review the trend of acute RV GE and acute GE admissions over the entire study period. | At least one year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Singapore, Singapore